CLINICAL TRIAL: NCT02703389
Title: Video, Ear Infections & Antibiotic Stewardship: Knowledge Translation Upon Emergency Department Discharge
Brief Title: Improving Knowledge Translation Upon Emergency Department Discharge
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Jeffrey Pernica, Head, Division of Pediatric Infectious Disease, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIF-2015-1123
Record Dates: First submitted 2016-03-02; First posted 2016-03-09 (Estimated); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Otitis Media
Keywords: knowledge translation; antimicrobial stewardship
MeSH Terms: conditions — Otitis Media | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Video (Experimental): An innovative video will be developed to explain the nature of non-severe acute otitis media and the rationale for watchful waiting and antimicrobial stewardship. This video will be viewed at recruitment and will be available online for further viewing later.
  Interventions: Behavioral: Video
- Pamphlet (Active Comparator): Informative pamphlet containing the same information as the video.
  Interventions: Behavioral: Pamphlet
- No intervention (No Intervention): This is the reference standard currently.

INTERVENTIONS:
Behavioral: Video — Animated video explaining acute otitis media and antimicrobial stewardship.
  Arms: Video
Behavioral: Pamphlet — Contains same information as video.
  Arms: Pamphlet

SUMMARY:
The amount and speed of emergency department (ED) discharge instructions often make it difficult for patients/caregivers to know the final diagnosis and to remember instructions. We hypothesize that a video on ear infections and antibiotics' role in their management will facilitate caregiver understanding and will increase the likelihood of caregivers properly following discharge instructions.

To verify this hypothesis, a large multi-centre clinical trial is needed. Prior to this, it is only ethical to conduct a smaller 'pilot' trial. Previously healthy children (6 months-5 years) diagnosed with mild ear infections at the McMaster Children's Hospital ED will be eligible to participate. If the child and caregiver decide to participate, before discharge, the caregiver will either: 1)watch the aforementioned video, 2)be given a pamphlet with the same information, or 3)standard of care (no additional information). Participants will fill a knowledge survey before discharge. The research assistant will contact all participants by phone to determine if the caregiver followed the discharge instructions.

DETAILED DESCRIPTION:
As most acute otitis media cases self-resolve, observation as initial management for mild acute otitis media (AOM) is recommended by Canadian and American authorities. However, North American children receive more antibiotics for AOM than for any other reason, making AOM-related prescribing a key focus for antimicrobial stewardship interventions. Low uptake of the ED suggested management strategies may be caused by caregiver under-appreciation of antibiotic-associated harms or from problems understanding the discharge plan, of which both could be remedied by a novel video-based knowledge translation platform.

The aim of this pilot study is to determine the feasibility of a follow-up large trial. The main clinical research question is: for caregivers of previously healthy children aged 6-59 months who are diagnosed by the ED physician with acute otitis media and judged to be eligible for a watchful waiting approach, will the use of an innovative informative video lead to lower rates of unnecessary antibiotic use as compared to a pamphlet or no intervention (reference standard)?

This will be a single-centre, randomized, controlled, pilot trial. Caregivers of previously well children aged 6-59 months presenting to the McMaster Children's Hospital (MCH) ED with non-severe AOM eligible for a watchful waiting approach will be enrolled and randomized to a video intervention, a pamphlet intervention, or standard care (no intervention). The primary outcome is the proportion of caregivers who fill a prescription for antimicrobials <48 hours after recruitment, as caregivers are generally advised to wait 48-72 hours prior to administering antibiotics to healthy children with mild AOM.

ELIGIBILITY:
Inclusion Criteria:

* caregivers of children aged 6-59 months diagnosed with non severe acute otitis media at the McMaster Children's Hospital ED

Exclusion Criteria:

* caregivers of children with severe symptoms (severe otalgia, fever > 39 C, impending perforation of tympanic membrane)
* caregivers who cannot readily access medical care
* caregivers who may not be able to recognize signs of worsening illness
* caregivers of children with immunodeficiency, malignancy, chronic cardiac or pulmonary disorders, anatomical abnormalities of head/neck, trisomy 21, or previous complicated otitis media

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 136 (Actual)
Dates: Start 2017-01; Primary Completion 2020-03 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who fill antimicrobial prescription early | <48 hours after recruitment
  The number of participants in each arm who fill and start administering a prescription for antimicrobials less than 48 hours after recruitment will be recorded.

SECONDARY OUTCOMES:
Proportion of participants who fill antimicrobial prescription inappropriately early | <48 hours after recruitment
  The number of participants in each arm who fill and start administering an 'inappropriate' prescription for antimicrobials - that is, if the child improves clinically - less than 48 hours after recruitment will be recorded.
Caregiver satisfaction with management plan (treatment arm) | 2-5 days after recruitment
  Caregiver satisfaction with the 'watchful waiting' strategy will be assessed using a Likert scale measure.
Caregiver retention of stewardship knowledge | 3 months after recruitment
  A quiz relating to antimicrobial stewardship will be administered at baseline and again at 3 months post-recruitment.

CONTACTS AND LOCATIONS:
Overall Officials: April Kam, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada